CLINICAL TRIAL: NCT01438931
Title: Phase III Randomized Placebo-controlled Double Blind Comparative Study to Investigate the Efficacy and Safety of DA-9501 in Sedation During the Surgery or Medical Procedure Without Intubation Under Monitored Sedation Care
Brief Title: Clinical Study to Investigate the Efficacy and the Safety of DA-9501 in Sedation During the Surgery or Medical Procedure Without Intubation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Maruishi Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEX-301
Record Dates: First submitted 2011-09-21; First posted 2011-09-22 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Sedation
Keywords: Dexmedetomidine; Sedation; Non-intubation; local anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo group (Placebo Comparator): Loading infusion of Placebo over 10 minutes followed by maintenance infusion of Placebo
  Interventions: Drug: placebo
- DA-9501 0.5 mcg/kg group (Active Comparator): Loading infusion of Dexmedetomidine 3.0 mcg/kg/hr over 10 minutes followed by maintenance infusion of Dexmedetomidine 0.2-0.7 mcg/kg/hr
  Interventions: Drug: DA-9501
- DA-9501 1.0 mcg/kg group (Active Comparator): Loading infusion of Dexmedetomidine 6.0 mcg/kg/hr over 10 minutes followed by maintenance infusion of Dexmedetomidine 0.2-0.7 mcg/kg/hr
  Interventions: Drug: DA-9501

INTERVENTIONS:
Drug: DA-9501 — Dexmedetomidine hydrochloride variable dose
  Arms: DA-9501 0.5 mcg/kg group; DA-9501 1.0 mcg/kg group
Drug: placebo
  Arms: Placebo group

SUMMARY:
The purpose of this study is to evaluate the efficacy and the safety of DA-9501 (Dexmedetomidine) in sedation during the surgery or medical procedure without intubation under monitored sedation care.

DETAILED DESCRIPTION:
Phase III, randomized, placebo controlled, double blind, parallel comparative study (Therapeutic confirmatory trial), to evaluate the efficacy and the safety of Dexmedetomidine in non-intubated patients who require sedation during surgery or medical procedure under monitored sedation care.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed and dated the Informed Consent after the study had been fully explained.
2. Patient is male or female, at least 20 years of age when the Informed Consent is obtained.
3. American Society for Anesthesiologists (ASA) I to III Class at the preoperative diagnosis.
4. New York Heart Association (NYHA) classification is I to III (Only patients who need classification of cardiac performance.)
5. Patient who requires sedation during the following elective surgery or procedure which require ≥30mins (expected time) without intubation under monitored sedation care.

   - Orthopedic, Otorhinologic, Oral surgeries, AV fistulas, Plastic, Excision of lesion, Breast biopsy, Catheter ablation, Vascular stents and AV shunt
6. Patient who requires local or regional anesthesia.

Exclusion Criteria:

1. Patient who underwent general anesthesia within 7 days, or who received other study drugs within 30 days from the date of consent.
2. Patient with <92% SpO2 at the physical examination prior to the study drug administration, or ventilatory failure which requires intubation or Laryngeal Mask.
3. Patient with central nervous system pathology which may lead to increased intracranial pressure, uncontrolled seizures, psychiatric disorder which may be confused with the response to sedation treatment.
4. Patient who require neurosurgical or cerebrovascular catheter procedures or interventions.
5. Patient who require general anesthesia, epidural anesthesia or spinal anesthesia for surgery or procedure.
6. Patient who receives treatment by alpha-2 agonists or alpha-2 antagonists within seven days of scheduled surgery or procedure.
7. Patient in whom opioids, DA-9501 or other alpha-2 agonists, or drugs which may be used in the study are contraindicated.
8. Patient diagnosed unstable angina or acute myocardiac infarction within 6 weeks from the date of consent.
9. Patient whose heart rate less than 50 bpm, systolic blood pressure less than 90 mm Hg by the physical examination prior to the study drug administration.
10. Patient has third degree heart block, unless the patient has a pacemaker.
11. Patient who has experienced an increase in alanine transaminase (ALT) and/or aspartate aminotransferase (AST) more than double the upper normal limit within 2 months of the date of consent, or who has a history of liver insufficiency.
12. Pregnant or lactating woman.
13. In the Investigator's or subinvestigator's opinion, patient has any symptom or factor, which might increase risk to the patient by conducting the study or preclude obtaining satisfactory study data.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Incidence of patients who did not require rescue administration of propofol to achieve and maintain Observer's Assessment of Alertness/Sedation (OAA/S) Score ≤4 during the study drug administration | Pre-dose, every 5 ± 2 minutes during study drug infusion and every 15 ± 2 minutes until 1 hour after study drug infusion. Before additional administration of sedative.

SECONDARY OUTCOMES:
Administration frequency and dosage of propofol required to achieve and maintain OAA/S score ≤4 during the study drug administration | After the start of study drug (20 ± 2 minutes), if the OAA/S score is 5.
  If the OAA/S score is 5, 0.2 mg/kg of propofol as a sedative is administered intravenously by slow "IV push" and the administration is to be repeated until the target level of sedation (OAA/S score ≤4) is achieved.
Time to first rescue administration of propofol | ≥15 minutes after the start of study drug infusion.
Incidence of patients who did not require rescue administration of fentanyl during the study drug administration | After the surgery start, the administration of fentanyl is permissible as required to treat pain. In case of repeated dose, the dosing interval should be ≥15 minutes.
Administration frequency and dosage of fentanyl required during the study drug administration | After the surgery start, the administration of fentanyl is permissible as required to treat pain. In case of repeated dose, the dosing interval should be ≥15 minutes.
Percentage of time spent OAA/S Score ≤4 during the study drug infusion | Pre-dose, every 5 ± 2 minutes during study drug infusion and every 15 ± 2 minutes until 1 hour after study drug infusion. Before additional administration of sedative.
Percentage of time spent OAA/S Score 3 to 4 during the study drug infusion | Pre-dose, every 5 ± 2 minutes during study drug infusion and every 15 ± 2 minutes until 1 hour after study drug infusion. Before additional administration of sedative.
Time to attain an Aldrete score ≥9 following discontinuation of the study drug infusion | Every 15 ± 2 minutes until the total score value becomes ≥9.
Visual Analogue Scale (VAS) score evaluation by Investigator or sub-investigator (ease of maintaining sedation level, hemodynamic stability, respiratory stability, subject's cooperativeness) | Within 24 hours after completion of the study drug administration
Score evaluation of satisfaction and anxiety of the subject | Within 24 hours after completion of the study drug administration (as much as possible)

CONTACTS AND LOCATIONS:
Locations (18):
- Japan (18):
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido
  - Hyogo Prefectural Amagasaki Hospital, Amagasaki, Hyōgo
  - Tsukuba University Hospital, Tsukuba, Ibaraki
  - Kagoshima University Medical and Dental Hospital, Kagoshima, Kagoshima-ken
  - Japanese Red Cross Kyoto Daini Hospital, Kyoto, Kyoto
  - University of Miyazaki Hospital, Miyazaki, Miyazaki
  - Okayama University Hospital, Okayama, Okayama-ken
  - Yuaikai Toyomijo Chuo Hospital, Toyomijo, Okinawa
  - Kansai Medical University Hirakata Hospital, Hirakata, Osaka
  - Kitano Hospital, The Tazuke Kofukai Medical Research Institute, Osaka, Osaka
  - Osaka Police Hospital, Osaka, Osaka
  - Osaka Saiseikai Nakatsu Hospital, Osaka, Osaka
  - Osaka University Dental Hospital, Suita, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Shimane University Hospital, Izumo, Shimane
  - Tottori University Hospital, Yonago, Tottori
  - Keio University Hospital, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo

REFERENCES:
- [Derived] Inagaki Y, Morita K, Ozaki M, Matsumoto K, Okayama A, Oya N, Hiraoka T, Takeda J. The Efficacy and Safety of Dexmedetomidine for Procedural Sedation in Patients Receiving Local Anesthesia Outside the Intensive Care Unit: A Prospective, Double-Blind, Randomized Clinical Phase III Trial in Japan. Yonago Acta Med. 2022 Jan 21;65(1):26-43. doi: 10.33160/yam.2022.02.005. eCollection 2022 Feb. PMID 35221758